CLINICAL TRIAL: NCT00183716
Title: An Randomized Controlled Trial (RCT) of the Trauma Recovery and Empowerment Model
Brief Title: The Trauma Recovery and Empowerment Model for Treating Post-Traumatic Stress Disorder in Women
Acronym: TREM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH068252 (NIH); R01MH068252 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Post-Traumatic Stress Disorder; Mental Disorders; Depression
Keywords: PTSD; Physical Abuse; Sexual Abuse; Women; Trauma; Group Therapy; Substance Abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Mental Disorders; Depression; Wounds and Injuries; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive Trauma Recovery and Empowerment Model and usual care
  Interventions: Behavioral: Trauma Recovery and Empowerment Model (TREM); Behavioral: Usual care
- 2 (Active Comparator): Participants will receive usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Trauma Recovery and Empowerment Model (TREM) — TREM is a 29-session group intervention for women who have experienced psychological trauma (e.g., childhood physical or sexual abuse), focusing on skill development, understanding the effects of trauma, and empowerment.
  Arms: 1
Behavioral: Usual care — Participants will receive usual care for women who have experienced psychological trauma.

SUMMARY:
This study will determine the effectiveness of the Trauma Recovery and Empowerment Model in reducing the severity of post-traumatic stress disorder symptoms in women with mental disorders and who have experienced sexual or physical abuse.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is an anxiety disorder that can develop after exposure to a terrifying event in which grave physical harm occurred or was threatened. Rates of PTSD are extremely high among people with severe mental disorders and such individuals find themselves at increased risk for depression, substance abuse, and poor overall health. In turn, these issues lead to high rates of utilization of mental health services. Unfortunately, there is currently a lack of effective trauma treatments that can be implemented in routine mental health settings. Trauma Recovery and Empowerment Model (TREM) is a group-based intervention that addresses PTSD and other closely related consequences of sexual and physical abuse among women with severe mental disorders. This study will determine the effectiveness of TREM in reducing the severity of PTSD symptoms in women with mental disorders who have experienced sexual or physical abuse.

Participants in this open label study will be randomly assigned to receive either usual care alone or usual care combined with TREM for 18 months. Usual care will include medication, case management, and therapy administered by a primary clinician. Participants assigned to usual care will report to the study site at least once a week, or as often as necessary. Participants assigned to usual care plus TREM will also be assigned to a primary clinician and will receive usual care as often as necessary. In addition, TREM participants will take part in 29 group sessions that will focus on increasing self-esteem and trauma-coping skills and reducing self-blame. PTSD symptom severity, trauma beliefs, depressive symptoms, substance use, and mental health service utilization will be measured at Months 6, 12, and 18 for all participants.

ELIGIBILITY:
Inclusion Criteria:

* History of physical and/or sexual abuse
* Diagnosis of a severe mental disorder
* Diagnosis of PTSD with a symptom severity score of 21 or higher

Exclusion Criteria:

* Severe developmental disabilities or organic brain damage

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
PTSD symptom severity | Measured at baseline and Months 6, 12, and 18

SECONDARY OUTCOMES:
Distorted beliefs | Measured at baseline and Months 6, 12, and 18
Depressive symptoms | Measured at baseline and Months 6, 12, and 18
Substance use | Measured at baseline and Months 6, 12, and 18
Mental health service utilization | Measured at Months 6, 12, and 18

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J. McHugo, PhD, Principal Investigator — Dartmouth College
Locations (2):
- United States (2):
  - Community Connections, Washington D.C., District of Columbia
  - The North Baltimore Center, Baltimore, Maryland